CLINICAL TRIAL: NCT04681911
Title: A Phase II Single-arm Clinical Trial of Inetetamab Combined With Pyrotinib and Chemotherapy in the Treatment of HER2 Positive Metastatic Breast Cancer
Brief Title: Inetetamab Combined With Pyrotinib and Chemotherapy in the Treatment of HER2 Positive Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jianli Zhao, Attending Doctor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-KY-125
Record Dates: First submitted 2020-10-25; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer
Keywords: HER2 positive metastatic breast cancer; Inetetamab; Pyrotinib
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Capecitabine; Gemcitabine; Vinorelbine; Carboplatin; Albumin-Bound Paclitaxel; eribulin

STUDY DESIGN:
Intervention Model Description: In order to improve the curative effect and prolong the survival rate, we added Inetetamab to the current second-line treatment regimen of Pyrotinib combined with chemotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inetetamab Combined With Pyrotinib and Chemotherapy (Experimental): Inetetamab: 8mg/kg for the first dose, 6mg/kg for the following doses, every 3 weeks for one cycle.
  Pyrotinib: 400mg, oral, every day.
  Chemotherapy: the choice of physicians，as the following regimens:
  Capecitabine, 1000 mg/m2, d1-d14, 3-week cycle Gemcitabine, 1000 mg/m2, D1, D8, 3-week cycle Vinorelbine, 25-30 mg/m2, D1, D8, 3-week cycle Carboplatin, AUC = 6, 3-week cycle Albumin paclitaxel, 100 mg/m2, weekly Eribulin, 1.4 mg/m2, D1, D8, 3-week cycle
  Interventions: Drug: Inetetamab; Drug: Pyrotinib; Drug: Capecitabine; Drug: Gemcitabine; Drug: Vinorelbine; Drug: Carboplatin; Drug: Albumin paclitaxel; Drug: Eribulin

INTERVENTIONS:
Drug: Inetetamab — Inetetamab: 8mg/kg for the first dose, 6mg/kg for the following doses, every 3 weeks for one cycle.
Drug: Pyrotinib — Pyrotinib: 400mg, oral, every day.
Drug: Capecitabine — Capecitabine, 1000 mg/m2, d1-d14, 3-week cycle
  Other Names: xeloda or other names
Drug: Gemcitabine — Gemcitabine, 1000 mg/m2, D1, D8, 3-week cycle
  Other Names: Gemzar or other names
Drug: Vinorelbine — Vinorelbine, 25-30 mg/m2, D1, D8, 3-week cycle
  Other Names: Navelbine or other names
Drug: Carboplatin — Carboplatin, AUC = 6, 3-week cycle
  Other Names: Paraplatin or other names
Drug: Albumin paclitaxel — Albumin paclitaxel, 100 mg/m2, weekly
  Other Names: Abraxane or other names
Drug: Eribulin — Eribulin, 1.4 mg/m2, D1, D8, 3-week cycle
  Other Names: Halaven

SUMMARY:
HER2-targeted therapy after the failure of trastuzumab treatment has become a new difficulty and challenge. Inetetamab, a new antibody to optimize the ADCC effect, has become one of the second-line treatment options after trastuzumab fails, showing good survival benefits. Pyrotinib, another second-line HER2 targeted drug, is a typical representative of TKI drugs, which not only has a strong HER2 antagonistic effect but also can synergize with monoclonal antibodies to amplify the ADCC effect. Pyrotinib and Inetetamab showed excellent anti-tumor efficacy and good safety in TKI and optimized ADCC respectively. we plan to carry out a phase II single-arm clinical study to evaluate the efficacy and safety of "Inetetamab combined with Pyrotinib and chemotherapy" in the treatment of her positive metastatic breast cancer.

DETAILED DESCRIPTION:
Trastuzumab is the first target drug for HER2 positive metastatic breast cancer, which can significantly improve the survival of patients with HER2 positive metastatic breast cancer and become the first-line standard treatment. However, the selection of second-line targeted drugs after the failure of trastuzumab treatment has become a new difficulty and challenge. Studies have shown that the ADCC effect is one of the main mechanisms of the anti-tumor effect of trastuzumab. Therefore, Inetetamab, a new antibody to optimize the ADCC effect, has become one of the second-line treatment options after trastuzumab fails, showing good survival benefits. Pyrotinib, another second-line HER2 targeted drug, is a typical representative of TKI drugs, which not only has a strong HER2 antagonistic effect but also can synergize with monoclonal antibodies to amplify the ADCC effect. As two important class 1.1 innovative drugs in China, Pyrotinib and Inetetamab showed excellent anti-tumor efficacy and good safety in TKI and optimized ADCC respectively. Considering that the current guidelines recommend the combination of multiple anti-HER2 targeted drugs, and basic research also shows that Pyrotinib and Inetetamab have a synergistic effect, we plan to carry out a phase II single-arm clinical study to evaluate the efficacy and safety of "Inetetamab combined with Pyrotinib and chemotherapy" in the treatment of her positive metastatic breast cancer, so as to provide better results for patients with HER2 positive metastatic breast cancer Treatment options!

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following conditions:

1. Adult female patients (age 18-70 years) with metastatic breast cancer confirmed by pathology or imaging;
2. Pathological diagnosis of HER-2 was positive (definition: immunohistochemical results were + + + or in situ hybridization results were positive);
3. Received trastuzumab treatment in the past;
4. the patients have received 1-3 treatments for metastatic breast cancer in the past;
5. According to RECIST 1.1, patients with at least one target lesion or simple bone metastasis can be evaluated;
6. ECoG score of physical status was less than 2, and the expected survival time was not less than 3 months;
7. Prior treatment-related toxicity should be reduced to NCI CTCAE (version 5.0) ≤ 1 degree (except for hair loss or other toxicity which is considered as no risk to patient's safety according to the investigator's judgment) 8）LVEF≥50%；

9) Sufficient functional reserve of bone marrow

1. White blood cell count (WBC) ≥ 3.0 × 10 ^ 9 / L,
2. Neutrophil count (ANC) ≥ 1.5 × 10 ^ 9 / L,
3. Platelet count (PLT) ≥ 100 × 10 ^ 9 / L 10) Previous treatment-related toxicity should be relieved as NCI CTCAE (version 5.0) ≤ 1 degree, total bilirubin (TBIL) ≤ 1.5 × upper limit of normal value (ULN), alanine aminotransferase (ALT / AST) ≤ 2.5 × ULN (liver metastasis patients ≤ 5xuln), serum creatinine ≤ 1.5 × ULN or creatinine clearance rate (CCR) ≥ 60 ml / min; 11) Be able to understand the research process, volunteer to participate in the study, and sign informed consent.

Exclusion Criteria:

Subjects were not allowed to participate in the study if they had any of the following conditions:

1. No trastuzumab treatment was received;
2. Have received more than 3 therapeutic regimens for metastatic breast cancer;
3. No treatment for metastatic breast cancer was received;
4. Patients who are known to be allergic to active or other components of the study drug.
5. They received radiotherapy, chemotherapy, endocrine therapy within 4 weeks before enrollment, or were participating in any clinical trials of intervention drugs;
6. Pregnant or lactating women, women of childbearing age who refused to take effective contraceptive measures during the study period.
7. Any other situation in which the researcher considers that the patient is not suitable for the study may interfere with the concomitant diseases or conditions involved in the study, or there are any serious medical barriers that may affect the safety of the subjects (e.g., uncontrollable heart disease, hypertension, active or uncontrollable infection, active hepatitis B virus infection)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2023-09-09 (Estimated); Study Completion 2024-09-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate，ORR | 18 weeks after enrollment
  Objective response rate assessed at 18 weeks after enrollment，that is about 6 cycles of treatment

SECONDARY OUTCOMES:
Progression Free Survival，PFS | 2 years
  The time from the beginning of treatment to the progression or death of the patient
overall survival，OS | 4 years
  The time from the beginning of treatment to the death of the patient
Clinical Benefit Rate，CBR | 24 weeks after enrollment
  Clinical Benefit Rate assessed at 24 weeks after enrollment，that is about 8 cycles of treatment
the rate of adverse events | up to 24 weeks after enrollment
  The probability and severity of adverse reactions were analyzed up to 24 weeks after enrollment
Quality of life scale score，QoL | 1 year
  The quality of life score of patients during treatment was analyzed（FACT-B）. Performance Status Rating (PSR) was demonstrated for the FACT-B total score, which is the result of the following subscale scores: SWB (the Social / family Well-Being subscale) , EWB (the Emotional Well-Being subscale), AC (Additional Concerns subscale), PWB (the Physical Well-Being subscale), FWB (the Functional Well-Being subscale)
Exploration of biomarkers | the first week after the enrollment
  Objective to explore the correlation between biomarkers and the ORR. The biomarkers will be test by nest-generation sequence, which include 520 genes and tumor mutation burden, like ERBB2/TP53/PIK3CA/ERBB4/CCND1 and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Jianli Zhao, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat Sen Memorial Hospital，Sun Yat sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
As personal information of patients is involved, we decided not to share individual participant data of patients.

REFERENCES:
- [Result] Li X, Yang C, Wan H, Zhang G, Feng J, Zhang L, Chen X, Zhong D, Lou L, Tao W, Zhang L. Discovery and development of pyrotinib: A novel irreversible EGFR/HER2 dual tyrosine kinase inhibitor with favorable safety profiles for the treatment of breast cancer. Eur J Pharm Sci. 2017 Dec 15;110:51-61. doi: 10.1016/j.ejps.2017.01.021. Epub 2017 Jan 21. PMID 28115222
- [Result] Ma F, Ouyang Q, Li W, Jiang Z, Tong Z, Liu Y, Li H, Yu S, Feng J, Wang S, Hu X, Zou J, Zhu X, Xu B. Pyrotinib or Lapatinib Combined With Capecitabine in HER2-Positive Metastatic Breast Cancer With Prior Taxanes, Anthracyclines, and/or Trastuzumab: A Randomized, Phase II Study. J Clin Oncol. 2019 Oct 10;37(29):2610-2619. doi: 10.1200/JCO.19.00108. Epub 2019 Aug 20. PMID 31430226
- [Result] Ma F, Li Q, Chen S, Zhu W, Fan Y, Wang J, Luo Y, Xing P, Lan B, Li M, Yi Z, Cai R, Yuan P, Zhang P, Li Q, Xu B. Phase I Study and Biomarker Analysis of Pyrotinib, a Novel Irreversible Pan-ErbB Receptor Tyrosine Kinase Inhibitor, in Patients With Human Epidermal Growth Factor Receptor 2-Positive Metastatic Breast Cancer. J Clin Oncol. 2017 Sep 20;35(27):3105-3112. doi: 10.1200/JCO.2016.69.6179. Epub 2017 May 12. PMID 28498781